CLINICAL TRIAL: NCT01828034
Title: A Phase I/II Study of First Line Gemcitabine, Cisplatin and MEK162 in Advanced Biliary Tract Carcinoma
Brief Title: First Line Gemcitabine, Cisplatin and MEK162 in Advanced Biliary Tract Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-004
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2019-06

CONDITIONS: Advanced Biliary Tract Carcinoma
Keywords: Gemcitabine; Cisplatin; MEK162; 13-004
MeSH Terms: interventions — Gemcitabine; Cisplatin; binimetinib

ARMS (1):
- Gemcitabine, Cisplatin and MEK162 (Experimental): Phase I component of the study, a classic 3+3 cohort dose escalation scheme will be used to identify the MTD of MEK162 when administered with gemcitabine at dose 800 mg/m2 and cisplatin given at dose 20 mg/m2 week 2 & 3 of a 3 week cycle. The final cohort will receive gemcitabine 1000mg/m2 and cisplatin 20mg/m2 week 2 and 3 of a 3 week cycle in combination with MEK162 at the MTD as determined above. In the phase II part of the study, patients will receive MEK162 at the MTD dose plus gemcitabine and cisplatin at the dose level determined acceptable in the phase I portion. In the phase II part of the study, patients will receive MEK162 at 45mg BID plus gemcitabine (800 mg/m2) and cisplatin (20 mg/m2) as determined by the phase I portion.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: MEK162

INTERVENTIONS:
Drug: Gemcitabine
Drug: Cisplatin
Drug: MEK162

SUMMARY:
The purpose of this study is to test an investigational combination of drugs for bile duct or gallbladder cancers. Gemcitabine and cisplatin are two forms of chemotherapy commonly used in combination to treat bile duct and gallbladder cancers. The investigators are looking to improve treatment results. They will attempt to do so by adding the drug MEK162 to the treatment plan. MEK162 acts by blocking a protein called MEK 1/2 which helps cancer cells grow and divide. This study will help answer the question of whether MEK162 is a helpful drug in patients with bile duct or gallbladder cancers when given with gemcitabine and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically / cytologically verified, non-resectable, recurrent, or metastatic biliary tract carcinoma including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder carcinoma. Combined cholangiocarcinoma and hepatocellular carcinoma is allowed.
* Patients must have measurable disease by RECIST 1.1
* KPS ≥ 80%
* Age ≥ 18 years
* Adequate bone marrow function defined as: Hb ≥ 8 g/dl, ANC ≥ 1.5 K/mcL, Platelets ≥ 100 K/mcL
* Adequate renal function defined as serum creatinine < 1.6 mg/dl and/or measured creatinine clearance from 24-hour urine collection of ≥ 60 ml/min
* Adequate hepatic function defined as total bilirubin ≤ 2 mg/dl, ALT/AST ≤ 5 x ULN.
* Patients with biliary obstruction can join if bilirubin corrects to required limit after adequate biliary drainage.

Adequate cardiac function defined as ejection fraction ≥ 45% as determined by transthoracic echocardiogram or MUGA

* Patients who have received prior local therapy, including but not limited to embolization, chemoembolization, radiofrequency ablation, radiation therapy, are eligible provided that measurable disease falls outside the treatment field or within the field but has shown an increase of ≥ 20% in the size. Prior local therapy must be completed at least 4 weeks prior to the baseline scan
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to study treatment
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any previous chemotherapy, biologic therapy, or investigational agent, except for adjuvant therapy as single agents and/or as radio-sensitizing agents limited to 5-fluorouracil and gemcitabine. Patient must have completed adjuvant therapy no less than six months prior to accrual.
* Evidence of another active cancer that may influence patient outcome as determined by the Principal Investigator (PI) or co-Principal Investigator (co-PI), except for nonmelanoma skin carcinoma, melanoma in-situ, in-situ carcinoma of the cervix curatively treated, treated superficial bladder cancer, and adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is non-detectable.
* Known brain metastases or primary central nervous system tumors with seizures that are not well controlled with standard medical therapy.
* Uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV positive patient
* Significant cardiovascular disease including congestive heart failure (New York Heart Association Class II or higher) or active angina pectoris.
* History of a myocardial infarction within 6 months.
* History of a stroke or transient ischemic attack within 6 months.
* Clinically significant peripheral vascular disease.
* Major surgical procedure within 4 weeks.
* Uncontrolled infection.
* Known or suspected allergy to gemcitabine or cisplatin
* Pregnant (positive pregnancy test)
* Breast-feeding should be discontinued if a nursing mother is to be treated on clinical trial.
* Any condition that impairs patient's ability to swallow whole pills
* Malabsorption problem that may limit or inhibit the absorption of MEK 162
* Patients with a history or current known evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or ophthalmopathy at baseline that would be considered a risk factor for CSR or RVO.
* History of any organ or bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Abou-Alfa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cohort 1
  Phase I, Dose Level 1 - MEK162 25 mg
- Cohort 2: Cohort 2 Phase I, Dose Level 2 - MEK162 45mg
- Cohort 3: Cohort 3 Phase I, Dose Level 3 / Phase II - MTD mg
- Cohort 4: Cohort 4 Phase II only, MTD mg
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 6 | 3 | 30
Completed | 3 | 6 | 3 | 29
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 29 | 41
Age, Continuous [Median (Full Range); unit: years] | 64.3 [56 to 72] | 54.3 [47 to 68] | 71.3 [69 to 76] | 69 [45 to 83] | 66 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 13 | 20
  Male | 1 | 3 | 1 | 16 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 3 | 27 | 37
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 2 | 5 | 2 | 27 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 3 | 29 | 41

OUTCOME MEASURES:

1. Primary Outcome: MTD of MEK162 - Phase I
Description: In the phase I portion, up to 18 patients will be enrolled in classic 3+3 cohort dose escalation design to identify the MTD of MEK162 when administered with gemcitabine and cisplatin given weeks 2 and 3 of a 3 week cycle .
Time Frame: 1 year
Measure: Number; unit: mg
Arm/Group | Gemcitabine, Cisplatin and MEK162
Number analyzed (Participants) | 12
mg | 45

2. Primary Outcome: Six-month Progression Free Survival
Description: An exact binomial single stage design will be used to discriminate between true 6-month PFS rates of 59% vs. 82%, and between true response rates of 26% and 50%. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Cisplatin and MEK162
Number analyzed (Participants) | 42
Participants
  Progression free | 19
  Progressed | 23

3. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: 1 participant withdrew consent before starting treatment
Measure: Number; unit: percentage of participants with ORR
Arm/Group | Gemcitabine, Cisplatin and MEK162
Number analyzed (Participants) | 41
percentage of participants with ORR | 12

4. Secondary Outcome: Median PFS
Description: progression free survival will be calculated from study entry to documented disease progression or death from any cause, whatever occurs first.
Time Frame: 1 year
Population: 1 participants withdrew consent before received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Cisplatin and MEK162
Number analyzed (Participants) | 41
months | 6 [4 to 12]

5. Secondary Outcome: Median Overall Survival
Description: (survival) will be calculated from study entry to death or last follow up
Time Frame: 1 year
Population: 1 participant withdrew consent before starting treatment
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Cisplatin and MEK162
Number analyzed (Participants) | 41
months | 13.3 [9.8 to 16.5]

6. Secondary Outcome: Participants Evaluated for Toxicity
Description: All toxicities will be rated as per the NCI Common Toxicity Criteria, version 4.
Time Frame: 2 years
Population: 1 participants withdrew consent before receiving treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Cisplatin and MEK162
Number analyzed (Participants) | 42
Participants
  Evaluated for toxicity | 41
  Not evaluable/withdrew consent before treatment | 1

ADVERSE EVENTS:
Time Frame: 2 years
Description: SAE's collected. Non-SAE/AE data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/6 | 1/3 | 16/29
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/6 | 3/3 | 29/29
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=3) | Cohort 4 (N=29)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 16
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 7
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7
Neutropenia (Investigations) | 1 | 1 | 2 | 20
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 17
Hyperlipasemia (Investigations) | 0 | 0 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT01828034/Prot_SAP_000.pdf